CLINICAL TRIAL: NCT04462133
Title: Optimal Tailored Treatment for H. Pylori Infection According to the Presence of DPO-PCR Based Clarithromycin Resistance
Brief Title: Optimal Tailored Treatment for H. Pylori Infection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study design was changed.
Sponsor: Incheon St.Mary's Hospital (Other)
Responsible Party: Principal Investigator, Joon Sung Kim, Assistant Proffessor, Incheon St.Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XC20ENDT0022
Record Dates: First submitted 2020-06-28; First posted 2020-07-08 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Helicobacter Pylori Infection; Antibiotic Resistant Infection

STUDY DESIGN:
Intervention Model Description: Empirical treatment versus tailored therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empirical therapy for H. pylori infection (Active Comparator): The empirical group receives triple therapy of 7 or 14 days for H. pylori eradication
  Interventions: Diagnostic Test: Dual-priming oligonucleotide-based multiplex polymerase chain reaction (DPO-PCR)
- Tailored therapy for H. pylori infection (Experimental): The tailored therapy group receives eradication regimens based on their DPO-PCR results. Triple therapy of 7 or 14 days for clarithromycin sensitive patients based on DPO-PCR and bismuth quadruple therapy of 7 or 14 days for clarithromycin resistant patients based on DPO-PCR.
  Interventions: Diagnostic Test: Dual-priming oligonucleotide-based multiplex polymerase chain reaction (DPO-PCR)

INTERVENTIONS:
Diagnostic Test: Dual-priming oligonucleotide-based multiplex polymerase chain reaction (DPO-PCR) — Empirical H. pylori eradication treatment versus tailored therapy based on DPO-PCR results

SUMMARY:
The efficacy of the current standard triple therapy is at an unacceptably low level. Resistance to antibiotics is suspected to be the major cause of the low efficacy of standard triple therapy. Point mutations in the 23S rRNA gene are known to be the primary mechanism of clarithromycin resistance against H pylori. Recently, a point mutation detection kit using a dual-priming oligonucleotide (DPO)-based multiplex polymerase chain reaction (PCR) assay was introduced and made commercially available. The primary goal of our study was to compare the eradication rates of empirical therapy and tailored therapy. Specifically we examined the eradication rates of 7-d, 14-d empirical therapy with 7-d, 14-d tailored therapy. Our secondary goal was to examine the adverse events of each treatment, cost effectiveness of each treatment methods, and accuracy of DPO-PCR for detecting H. pylori resistance.

DETAILED DESCRIPTION:
Patients are randomly assigned to the empirical therapy group and tailored therapy group.

The empirical therapy group recieves triple therapy of 7 or 14 days. The tailored therapy group receives treatment based on their DPO-PCR results.

Patients who are sensitive to clarithromycin based on DPO-PCR receives triple therapy for 7 or 14 days. Patients who are resistant to clarithromycin based on DPO-PCR recieves bismuth quadruple therapy for 7 or 14 days.

ELIGIBILITY:
Inclusion Criteria:

* consecutive subjects who underwent upper gastrointestinal endoscopy and who had a confirmed diagnosis of H pylori infection

Exclusion Criteria:

* subjects younger than 18 years old
* subjects with a history of H pylori eradication
* subjects who had previous gastric surgery
* subjects who were pregnant or lactating
* subjects with serious concurrent illness
* subjects who were administered antibiotics, bismuth, or PPIs in the 8 weeks preceding the study
* subjects with a history of allergy to any one of the compounds in this study

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Eradication success | 8-12 weeks after eradication
  H. pylori eradication success based on urea breath test

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Wook Kim, MD, PhD, Principal Investigator — Incheon St.Mary's Hospital
Locations (1):
- Incheon St. Mary's Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No